CLINICAL TRIAL: NCT07401316
Title: Circulating Tumor DNA in Stage I, II, and III Germ-Cell Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Principal Investigator, Nabil Adra, Associate Professor of Clinical Medicine, Indiana University
Other Study IDs: CTO-IUSCCC-0937
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Germ Cell Cancer Metastatic
Keywords: ctDNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Cohort I - High Risk Clinical stage I: 50 subjects will be enrolled with high-risk stage I seminomatous or non-seminomatous germ cell tumors. In these patients, ctDNA will be collected post-orchiectomy prior to initiation of surveillance and every 4 months during surveillance for up to 2 years.
  Interventions: Diagnostic Test: Whole blood for ctDNA
- Cohort II- Clinical stage II: 30 patients will be enrolled with clinical Stage II seminomatous or non-seminomatous germ cell tumor who are planning to undergo primary resection with RPLND. In these patients, ctDNA will be collected prior to surgery and every 4 months after surgery for up to 2 years.
  Interventions: Diagnostic Test: Whole blood for ctDNA
- Cohort III- Clinical stage III: 50 patients will be enrolled with clinical Stage III (or IS) seminomatous or non-seminomatous germ cell tumor who are planning to undergo first-line chemotherapy. In these patients, ctDNA will be collected prior to chemotherapy, at cycle 2 day 1, and every 4 months after completing chemotherapy.
  Interventions: Diagnostic Test: Whole blood for ctDNA

INTERVENTIONS:
Diagnostic Test: Whole blood for ctDNA — Whole blood for ctDNA

SUMMARY:
This study will evaluate the utility of ctDNA detection in patients with high-risk stage I, stage II, and stage III germ cell tumor disease to develop a tool for post-treatment cancer cell detection.

DETAILED DESCRIPTION:
This is a specimen collection study where patients with high-risk stage I germ cell tumor, clinical stage II germ cell tumor, and clinical stage III germ cell tumor will be evaluated for ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Subjects must have histologically or serologically confirmed seminomatous or non seminomatous germ cell tumor. Non-seminoma includes embryonal carcinoma, choriocarcinoma, yolk sac tumor, or teratoma.

   Note: Cohort I is for high-risk clinical stage I disease. Cohort II is for clinical stage II. Cohort III is for clinical stage III or IS.
4. Archival tissue for germ-cell tumor diagnosis available

Exclusion Criteria:

1. Concurrent disease or condition that would make the subject inappropriate for study participation
2. Any serious medical disorder that would interfere with the subject's safety
3. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent per treating physician coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients have been diagnosed with either high-risk stage I or clinical stage II germ cell tumors (GCT) and are planning to receive standard of care (SOC) treatment; including either an orchiectomy (a surgical procedure that removes one or both testicles) for stage I, or a retroperitoneal lymph node dissection (RPLND) (surgery to remove the lymph nodes in the back of the abdomen).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value (PPV) of circulating tumor DNA in Cohort I | At screening and every 4 months up to 2 years
  PPV will be calculated as the number of true positives divided by the total number of positive tests in patients with high-risk stage I germ cell tumor.
Positive predictive value (PPV) of circulating tumor DNA in Cohort II | At screening and every 4 months up to 2 years
  PPV will be calculated as the number of true positives divided by the total number of positive tests in the node dissection patients with clinical stage II germ cell tumor.
Positive predictive value (PPV) of circulating tumor DNA in Cohort III | At screening and every 4 months up to 2 years
  PPV will be calculated as the number of true positives divided by the total number of positive tests in the first-line chemotherapy patients with clinical stage III germ cell tumor.

SECONDARY OUTCOMES:
Negative predictive value (NPV) of circulating tumor DNA in Cohort I | At screening and every 4 months up to 2 years
  NPV will be calculated as the number of true negatives divided by the total number of negative tests in patients with high-risk stage I germ cell tumor.
Negative predictive value (NPV) of circulating tumor DNA in Cohort II | At screening and every 4 months up to 2 years
  NPV will be calculated as the number of true negatives divided by the total number of negative tests in the node dissection patients with clinical stage II germ cell tumor.
Negative predictive value (NPV) of circulating tumor DNA in Cohort III | At screening and every 4 months up to 2 years
  NPV will be calculated as the number of true positives divided by the total number of positive tests in the first-line chemotherapy patients with clinical stage III germ cell tumor.
Post-node dissection circulating tumor DNA bioassay | At screening and every 4 months up to 2 years
  Means/stds of ctDNA in both the relapsed and non-relapsed patients in Cohort II.
Post-node dissection clearance rate of ctDNA | At screening and every 4 months up to 2 years
  The clearance rate of ctDNA in the node dissection patients in Cohort II.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Adra, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States